CLINICAL TRIAL: NCT06508047
Title: Respiratory Rate Validation Study - Mindset Medical Informed Vital Core Application
Status: Completed | Type: Observational
Sponsor: Mindset Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: PR 2024-593
Record Dates: First submitted 2024-07-12; First posted 2024-07-18 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Vital Sign Evaluation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Informed Vital Core App: All subjects assigned to a single arm, respiration rate measurement will be collected, calculated, and displayed on the web based application. Conventional Capnography will also be used to collect and display the respiratory rate at the same time as the Informed Vital Core App.
  Interventions: Device: Informed Vital Core App

INTERVENTIONS:
Device: Informed Vital Core App — Informed Vital Core App will be initiated by the study staff to take a measurement, which takes 60 seconds to calculate and report a breathing rate value.

SUMMARY:
Evaluating the Accuracy of a Web-Based Application - Vital Sign Measurement Platform. This single-arm cohort, open-label study is designed to evaluate the accuracy of a web-based application designed for measurements of vital signs including respiratory rate (RR). The purpose of the study is to conduct accuracy validation when compared to a FDA-cleared/approved vital sign monitoring device (reference device).

ELIGIBILITY:
Inclusion Criteria:

* Participants must have the ability to understand and provide written informed consent or have legally authorized representative consent to participate.
* Participant must be ≥22 years of age
* Participant must be willing and able to comply with study procedures and duration
* Participants or legally authorized representative must be able to read or write in English

Exclusion Criteria:

* Participants who refuse or are unable to sign an informed written consent for study
* Participants evaluated by the Investigator and Clinical Staff and found to be medically unsuitable or have self-reported health conditions that are currently unstable as identified in the Health Assessment Form and Health Screening
* Compromised circulation, injury, or physical malformation the Region of Interest (ROI) which would limit the ability to test ROI needed for the study. (Note: Certain malformations may still allow participants to participate if the condition is noted and would not affect the particular areas utilized.)
* Participants with severe contact allergies to standard adhesives, latex or other materials found in pulse oximetry sensors, ECG electrodes, or other medical sensors (self-reported)
* Other known health condition, should be considered upon disclosure in health assessment form

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: At least 30% of the participants will be male At least 30% of the participants will be female
  At least 33% of the participants will be with BMI between 25.0 to 29.9 kg/m2 (overweight) At least 33% of the participants will be with BMI > 30.0 kg/m2 (obese)
  At least 15% of participants will have a light skin tone (Fitzpatrick Scale 1 or 2) At least 15% of participants will have a medium skin tone (Fitzpatrick Scale 3 or 4) At least 15% of participants will have a dark skin tone (Fitzpatrick Scale 5 or 6)
  The study will attempt to enroll a race/ethnicity distribution similar to population demographics consistent with the 2020 US Census Data
  At least 5 participants will have a history of smoking
  At least 10 participants with chronic conditions (self-reported):
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2024-07-16 (Actual); Primary Completion 2024-08-22 (Actual); Study Completion 2024-08-22 (Actual)

PRIMARY OUTCOMES:
Respiratory Rate Accuracy | 60 seconds
  The primary outcome measure is a Respiratory Rate accuracy validation comparing the Mindset Medical Application to the Reference, an FDA cleared End Tidal Carbon Dioxide monitor (GE Datex-Ohmeda) by manually scoring the collected waveform for data analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Monica Rabanal, Principal Investigator — Element Materials Technology
Locations (1):
- Element Materials Techonology, Louisville, Colorado, United States

IPD SHARING:
Plan to Share IPD: No